CLINICAL TRIAL: NCT01052844
Title: Clinical Trial of Gabapentin in the Prevention of Nausea Ond Vomiting Induced by Chemotherapy, a Randomized, Double-blind, Placebo Controled Study
Brief Title: Gabapentin in the Prevention of Nausea and Vomiting Induced by Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Felipe Melo Cruz, MsC, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABC-2009
Record Dates: First submitted 2009-12-17; First posted 2010-01-20 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-01

CONDITIONS: Vomiting; Cisplatin Adverse Reaction
Keywords: Vomiting; Antiemetics; Dexamethasone; Cisplatin; Antineoplastic combined chemotherapy protocols
MeSH Terms: conditions — Vomiting | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): Placebo:
  * Five and four days before chemotherapy (day -5 and day -4): 1x daily
  * Three and two days before chemotherapy (day -3 and day -2): 2x daily
  * One day before to five days after chemotherapy ( day -1 to day 5): 3x daily
  Interventions: Drug: Placebo
- Gabapentin (Experimental): Gabapentin 300mg:
  * Five and four days before chemotherapy (day -5 and day -4): 1x daily
  * Three and two days before chemotherapy (day -3 and day -2): 2x daily
  * One day before to five days after chemotherapy ( day -1 to day 5): 3x daily
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Placebo — Placebo, given orally Ranitide 50 mg, IV, before chemotherapy (D1) Ondansetron 8 mg, IV, before chemotherapy (D1) Dexamethasone 10 mg, IV, before chemotherapy (D1) Dexamethasone 4 mg, PO, 2x/day (D2, D3)
  Arms: Control group
Drug: Gabapentin — Gabapentin 300mg, orally Ranitide 50 mg, IV, before chemotherapy (D1) Ondansetron 8 mg, IV, before chemotherapy (D1) Dexamethasone 10 mg, IV, before chemotherapy (D1) Dexamethasone 4 mg, PO, 2x/day (D2, D3)
  Arms: Gabapentin

SUMMARY:
Gabapentin is an antiepileptic drug. Its antiemetic effect is demonstrated after laparoscopic surgery, but it is not yet known whether gabapentin is effective in preventing chemotherapy induced emesis.

The purpose of this study is to determine whether the addition of gabapentin to dexamethasone plus ondansetron increase the control of chemotherapy-induced nausea and vomiting.

DETAILED DESCRIPTION:
This was a prospective, double-blind, placebo-controlled study conducted at our institution (Faculdade de Medicina da Fundação ABC and affiliated Hospitals) from April 2009 to April 2010. Patients and personnel involved in the study were blinded to the assigned treatment. The study was approved by the ethics committee of our institution. All the patients provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* First course of chemotherapy ( cisplatin or doxorubicin at a dose of at least 50mg per square meter)
* Written informed consent must be obtained before initiating the protocol procedures

Exclusion Criteria:

* ECOG 3
* Nausea and vomiting within the past 1 day
* Gastrointestinal obstruction
* Concurrent use of opioid
* Patients with brain metastases
* History of allergic or other adverse reaction to gabapentin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Auro del Giglio, phD, Study Director — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil

REFERENCES:
- [Derived] Cruz FM, de Iracema Gomes Cubero D, Taranto P, Lerner T, Lera AT, da Costa Miranda M, da Cunha Vieira M, de Souza Fede AB, Schindler F, Carrasco MM, de Afonseca SO, Pinczowski H, del Giglio A. Gabapentin for the prevention of chemotherapy- induced nausea and vomiting: a pilot study. Support Care Cancer. 2012 Mar;20(3):601-6. doi: 10.1007/s00520-011-1138-4. Epub 2011 Apr 5. PMID 21465325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, double-blind, placebo-controlled study conducted at our institution (Faculdade de Medicina da Fundação ABC and affiliated Hospitals) from April 2009 to April 2010. Patients and personnel involved in the study were blinded to the assigned treatment.
Pre-assignment Details: Patients and personnel involved in the study were blinded to the assigned treatment. The study was approved by the ethics committee of our institution. All the patients provided written informed consent. No enrolled participants were excluded from the trial.
Groups:
- Control Group: Dexamethasone 10mg + Ondansetron 8mg + Ranitidine 50mg , IV, before chemotherapy infusion (D1)
  Dexamethasone 8mg orally 24h (day 2) and 48h (day 3) after chemotherapy
  Placebo:
  * Five and four days before chemotherapy (day -5 and day -4): 1x daily
  * Three and two days before chemotherapy (day -3 and day -2): 2x daily
  * One day before to five days after chemotherapy ( day -1 to day 5): 3x daily
- Gabapentin: Dexamethasone 10mg + Ondansetron 8mg + Ranitidine 50mg , IV, before chemotherapy infusion (D1)
  Dexamethasone 8mg orally 24h (day 2) and 48h (day 3) after chemotherapy
  Gabapentin 300mg:
  * Five and four days before chemotherapy (day -5 and day -4): 1x daily
  * Three and two days before chemotherapy (day -3 and day -2): 2x daily
  * One day before to five days after chemotherapy ( day -1 to day 5): 3x daily
Period: Overall Study
Arm/Group | Control Group | Gabapentin
Started | 40 | 40
Completed | 40 | 39
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Gabapentin | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 34 | 68
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (10.4) | 55.6 (9.9) | 53.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 75
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  Brazil | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Response During Chemotherapy Course 1
Description: The CR was defined as no emetic episodes and no nausea episodes from day 1 to day 5 (0-120h)
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Control Group | Gabapentin
Number analyzed (Participants) | 40 | 40
participants | 17 | 26
Statistical Analysis 1: Comparison: Control Group vs Gabapentin; Complete protection from nausea and vomiting (CP) was defined as the absence of any episode of nausea or vomiting and no use of rescue medication. CP was further defined as either acute (ACP), when occurring during the first 24 hours after chemotherapy; delayed (DCP), when occurring during the period from days 2 through 5 after chemotherapy; or overall, when occurring over the entire period of the study (first 120 hours); Test type: Superiority or Other; p = 0.04, Chi-squared

2. Primary Outcome: Number of Patients With CR During Delayed-onset Phase (24-120 Hours) After Administration of Chemotherapy Course 1
Description: Complete response during delayed-onset phase was defined as the absence of any episode of nausea or vomiting and no use of rescue medication when occurring during the period from days 2 through 5 after chemotherapy
Time Frame: 6 days
Measure: Number; unit: participants
Arm/Group | Control Group | Gabapentin
Number analyzed (Participants) | 40 | 40
participants | 21 | 29
Statistical Analysis 1: Comparison: Control Group vs Gabapentin; We evaluated associations between categorical variables using the Chi-Square test; Test type: Superiority or Other; p = 0.06, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data were colected from day 1 to day 6 after chemotherapy
Arm/Group | Control Group | Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 22/40 | 23/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=40) | Gabapentin (N=40)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Constipation (Gastrointestinal disorders) | 12 (12) | 18 (18)
Xerostomia (Gastrointestinal disorders) | 19 (19) | 23 (23)
Heartburn (Gastrointestinal disorders) | 10 (10) | 13 (13)
Sleepiness (Nervous system disorders) | 19 (19) | 18 (18)
Dizziness (Ear and labyrinth disorders) | 13 (13) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No